## STATISTICAL ANALYSIS PLAN

#### CCD-5633AA1-02

ClinicalTrials.gov ID: NCT02452476

A MULTICENTER, DOUBLE BLIND, RANDOMIZED, SINGLE DOSE, ACTIVE-CONTROLLED STUDY TO INVESTIGATE THE EFFICACY AND SAFETY OF SYNTHETIC SURFACTANT (CHF 5633) IN COMPARISON TO PORCINE SURFACTANT (PORACTANT ALFA, CUROSURF®) IN THE TREATMENT OF PRETERM NEONATES WITH RESPIRATORY DISTRESS SYNDROME.

Version: Final 1.0

Date: 18/Jul/2018

Chiesi Final 1.0 CCD-5633AA1-02 18/July/2018

TP-EP.BS-WW-001-05 Effective date: 29 Jul 15

Related to: SOP-EP.BS-WW-002 



# **REVISION HISTORY**

| Version | Version Date | Author | <b>Summary of Changes Made</b> |
|---|---|---|---|
| Draft 0.1 | 07/Dec/2015 | | New Document |
| Draft 0.2 | 03/Feb/2016 | | Implementation of sponsor comments |
| Draft 0.3 | 24/Feb/2016 | | Incorporated sponsor comments plus refinements. |
| Draft 0.4 | 17/Mar/2016 | | Incorporated sponsor comments and display of protocol deviations and screening failures |
| Draft 0.5 | 15/Apr/2016 | | Incorporated sponsor comments |
| Draft 0.6 | 09/May/2018 | | Updates for Protocol Amendment 4.0 (dated 31/Jan/2018) and sponsor comments |
| Draft 0.7 | 29/May/2018 | | Implementation of sponsor comments |
| Draft 0.8 | 27/Jun/2018 | | Implementation of sponsor comments |
| Draft 0.9 | 13/Jul/2018 | | Implementation of sponsor comments |
| Final 1.0 | 18/Jul/2018 | | Comments resolution |

Chiesi Final 1.0 CCD-5633AA1-02 18/July/2018

TP-EP.BS-WW-001-05 Effective date: 29 Jul 15

Related to: SOP-EP.BS-WW-002 

# TABLE OF CONTENTS

| REVIS | SION HI | ISTORY | | 2 |
|---|---|---|---|---|
| TABL | E OF C | ONTEN | TS | 3 |
| LIST ( | OF IN-T | EXT TA | BLES / FIGURES | 5 |
| ABBR | EVIAT | ION AN | D ACRONYM LIST | 6 |
| STATI | [STICA] | L ANAL | YSIS PLAN | 9 |
| 1. | STUD | Y OBJE | CTIVES | 9 |
| | 1.1 | Primar | ry Objectives | 9 |
| | 1.2 | | lary Objectives | |
| 2. | STUDY DESIGN | | | |
| 3. | STUD | Y POPU | ILATION | 10 |
| 4. | | | _ BASIS FOR SAMPLE SIZE | |
| 5. | | | TION | |
| 6. | | | L ANALYSIS CONVENTIONS | |
| 0. | 6.1 | | ted Data | |
| | 0.1 | 6.1.1 | Disposition data | |
| | | 6.1.2 | Demographic and Background Data | |
| | | 6.1.3 | Safety Data | |
| | | | 6.1.3.1 Adverse Events and Adverse Drug Reactions | |
| | | | 6.1.3.2 Clinical Laboratory Tests | |
| | | | 6.1.3.3 Vital Signs | |
| | | | 6.1.3.4 Physical Examination | |
| | | | 6.1.3.6 Surgical/ Medical Procedures | |
| | | | 6.1.3.7 Immunogenicity Assessment | |
| | | 6.1.4 | Pharmacodynamic/Efficacy Data | |
| | | | 6.1.4.1 Ratio of arterial oxygen saturation (SpO <sub>2</sub> /FiO <sub>2</sub> ) | |
| | | | 6.1.4.2 Fraction of inspired oxygen (FiO <sub>2</sub> ) | |
| | | | 6.1.4.3 Arterial oxygen saturation (SpO2) | |
| | | | 6.1.4.4 Respiratory Severity Score (RSS) | |
| | | | 6.1.4.5 Oxygen Saturation Index (OSI) | 19 |
| | | | 6.1.4.6 Ventilator Settings | |
| | | | 6.1.4.7 Biomarkers of inflammation | |
| | | | 6.1.4.9 Rescue medication | |
| | | | 6.1.4.10 Respiratory Support and Related Duration of Ventila | |
| | | | and Non-invasive) | |
| | | | 6.1.4.11 Oxygen Use and Related Duration | |
| | | | 6.1.4.12 Normal breathing (i.e. at room air) patients within 24 | |
| | | | 6.1.4.13 Alveolar–Arterial Gradient | |
| | | | 6.1.4.14 Oxygenation Index | |
| Chiesi | | | | Final 1.0 |
| | -5633A | <b>41-02</b> | | 18/July/2018 |
| - | | | | J |

TP-EP.BS-WW-001-05 Effective date: 29 Jul 15

Related to: SOP-EP.BS-WW-002 

| | 6.2 | Analys | is Populat | ions | 24 |
|---|---|---|---|---|---|
| | | 6.2.1 | Safety Po | opulation | 24 |
| | | 6.2.2 | | i-to-Treat Population | |
| | | 6.2.3 | | ocol Population | |
| | 6.3 | Statistic | | sis Methods | |
| | 0.0 | 6.3.1 | • | and Descriptive Statistics | |
| | | 6.3.2 | | Il Significance Level | |
| | | 6.3.3 | | Significance Level | |
| | | 6.3.4 | | Data | |
| | | 6.3.5 | _ | Analysis | |
| | | 6.3.6 | | Deviations | |
| | | 6.3.7 | | disposition | |
| | | 6.3.8 | | aphic Data | |
| | | 6.3.9 | | and Neonatal Concomitant Medication | |
| | | 6.3.10 | | e to the Investigational Medicinal Product | |
| | | 6.3.11 | | nalysis | |
| | | 0.5.11 | | Adverse Events | |
| | | | | Clinical Safety Laboratory Tests (hematology, biochemistry) | |
| | | | | Vital Signs | |
| | | | | Immunogenicity data | |
| | | 6.3.12 | | Variables | |
| | | 0.0.12 | • | Statistical Analysis | |
| | | 6.3.12.1 | | SpO <sub>2</sub> /FiO <sub>2</sub> Ratio | |
| | | 6.3.12.1 | | FiO2 | |
| | | 6.3.12.1 | | RSS | |
| | | 6.3.12.1 | | OSI | |
| | | 6.3.12.1 | | SpO2 | |
| | | 6.3.12.1 | | Ventilator Settings | |
| | | 6.3.12.1 | | BPD incidence, Mortality/BPD incidence, mortality and I | |
| | | | mortality | · | |
| | | 6.3.12.1 | .8 | Rescue surfactant use | 34 |
| | | 6.3.12.1 | .9 | Duration of ventilation and oxygen use | 34 |
| | | 6.3.12.1 | .10 | Normal breathing patients within 24 hours | 35 |
| | | 6.3.12.1 | .11 | Biomarkers of inflammation | 35 |
| | | 6.3.12.1 | .12 | Alveolar-Arterial Gradient | 36 |
| 7. | REFER | RENCES | | | 37 |
| 8. | | | | GS TO BE INCLUDED IN SECTION 14 OF THE CLINI | |
| 8. | | | | 55 TO BE INCLUDED IN SECTION 14 OF THE CLINIC | |
| 9. | | | | CLUDED IN SECTION 16 OF THE CLINICAL STU | |
| 10. | DOCU | MENTA | TION OI | STATISTICAL METHODS | 44 |
| 11. | | | | | |
| 11. | | | | | |
| | 11.1 | Study S | scnedule ( | according to protocol Amendment 1) | 45 |
| C1 : : | | | | | D' 110 |
| Chiesi | | | | | Final 1.0 |

TP-EP.BS-WW-001-05 Effective date: 29 Jul 15

CCD-5633AA1-02

Related to: SOP-EP.BS-WW-002 

18/July/2018

## LIST OF IN-TEXT TABLES / FIGURES

Not applicable.

Chiesi Final 1.0 CCD-5633AA1-02 18/July/2018

TP-EP.BS-WW-001-05 Effective date: 29 Jul 15

Related to: SOP-EP.BS-WW-002 

## ABBREVIATION AND ACRONYM LIST

## Abbreviation / Acronym Definition / Expansion

ADR Adverse drug reactions

AE Adverse event

ALT alanine aminotransferase
AOP Apnea of prematurity

AST aspartate aminotransferase

ATC Anatomical therapeutic chemical
BiPAP Bi-level positive airway pressure
BPD Bronchopulmonary dysplasia

bpm Beats per minute
CI Confidence interval

CMH Cochran-Mantel-Haenszel

CPAP Continuous Positive Airway Pressure

CS Clinically significant or Cranial Sonography

CSP Clinical Study Protocol

CX Chest X-Ray

DBP Diastolic blood pressure

eCRF Electronic Case Report Form

FBC Full blood count

FiO<sub>2</sub> Fraction of inspired oxygen

GA Gestational age
GMH Germinal matrix

H High (value above upper limit of reference range)

HFNC High flow nasal cannula

HFOV High Frequency Oscillatory Ventilation

HL Hodges-Lehmann

HR Heart rate

IL1β Interleukin 1β

Chiesi Final 1.0

CCD-5633AA1-02

TP-EP.BS-WW-001-05 Effective date: 29 Jul 15

Related to: SOP-EP.BS-WW-002 

Abbreviation / Acronym Definition / Expansion

IL6 Interleukin 6

IMV Intermittent Mandatory Ventilation

IRT Interactive Response Technology

ITT Intention to treat (population)
IVH Intraventricular hemorrhage

IVRS Interactive Voice Response Services
IWRS Interactive Web Response System

Low (value below lower limit of reference range)

MAP Mean airway pressure

MedDRA Medical Dictionary for Regulatory Activities

MMRM Mixed model for repeated measures

MOP Myeloperoxidase

NC Neonatal Complications of prematurity

NCS Not clinically significant
NEC Necrotizing enterocolitis

NHFV Nasal High frequency ventilation

nIMV Nasal Intermittent Mandatory Ventilation

NIPPV Nasal intermittent positive pressure ventilation

NK Not known

NPSV Nasal Pressure Support Ventilation

nSIMV Nasal Synchronized Intermittent Mandatory Ventilation

nSIPPV Nasal Synchronized Intermittent Positive Pressure Ventilation

OI Oxygenation index

OR Odds ratio

OSI Oxygen saturation index

PaO<sub>2</sub> Partial pressure of oxygen in arterial blood

PDA Patent ductus arteriosus

PEEP Positive end-expiratory pressure

PH Pregnancy history

Chiesi Final 1.0

CCD-5633AA1-02

TP-EP.BS-WW-001-05 Effective date: 29 Jul 15

Related to: SOP-EP.BS-WW-002 

## Abbreviation / Acronym Definition / Expansion

PIE Pulmonary interstitial emphysema

PIP Peak inspiratory pressure

PK Pharmacokinetic

PMA post menstrual age

PNA post-natal age

POC Proof of Concept

PP Per protocol

PT Preferred term

PTV Patient trigger ventilation

PVL Periventricular leukomalacia

RDS Respiratory Distress Syndrome

ROP Retinopathy of prematurity

RR Relative risk

RSS Respiratory severity score

SAE Serious adverse event

SAF Safety Population

SAP Statistical Analysis Plan

SBP Systolic blood pressure

SD Standard deviation or single dose

SE Standard error

SIMV Synchronized intermittent mandatory ventilation

SIPPV Synchronized intermittent positive pressure ventilation

SOC System Organ Class

SpO<sub>2</sub> Arterial oxygen saturation

TEAE Treatment-emergent adverse event

TLF Tables, Listings and Figures

TNF-α Tumor Necrosis Factor-alpha

VS Ventilatory Support

WHO-DD World Health Organization - Drug Dictionary

Y/N Yes/No

Chiesi Final 1.0

CCD-5633AA1-02 18/July/2018

TP-EP.BS-WW-001-05 Effective date: 29 Jul 15

Related to: SOP-EP.BS-WW-002

#### STATISTICAL ANALYSIS PLAN

The Statistical Analysis Plan (SAP) details the statistical methodology to be used in analyzing study data and outlines the statistical programming specifications for the Tables, Listings and Figures (TLFs). It describes the variables and populations, anticipated data transformations and manipulations and other details of the analyses not provided in the Clinical Study Protocol (CSP).

The analyses described are based on the final amended CSP Version 4.0, dated, 31/Jan/2018.

The SAP will be finalized prior to database lock and describes the statistical analysis as it is foreseen when the study is being planned. If circumstances should arise during the study rendering this analysis inappropriate, or if improved methods of analysis should arise, updates to the analyses may be made. Any deviations from the SAP after database lock, reasons for such deviations and all alternative or additional statistical analyses that may be performed, will be described in a SAP Addendum.

The 24-months assessment analysis will be described in a separate SAP.

#### 1. STUDY OBJECTIVES

This trial is a multicenter, double-blind, randomized, single dose, active-controlled, Proof of Concept (POC)/Phase II study to investigate the efficacy and safety of synthetic surfactant (CHF 5633) in comparison to porcine surfactant (Poractant alfa, Curosurf ®) in the treatment of preterm neonates with Respiratory Distress Syndrome (RDS).

## 1.1 Primary Objectives

Main objectives of this study are:

- to investigate the short term efficacy profile of CHF 5633 vs. porcine surfactant (Poractant Alfa, Curosurf®) in terms of reduced oxygen requirement and ventilatory support (VS)
- to evaluate the mid-term efficacy profile in terms of reduced incidence of bronchopulmonary dysplasia (BPD) and mortality/BPD rate at 36 weeks post menstrual age (PMA), mortality rate at 28 days post-natal age (PNA) and 36 weeks PMA, RDS-associated mortality through 14 days of age and other major co-morbidities of prematurity.

#### 1.2 Secondary Objectives

Other objectives of the present study are:

Chiesi Final 1.0

CCD-5633AA1-02 18/July/2018

- to evaluate the need for re-dosing in the two treatment groups according the pre-defined criteria;
- to evaluate the inflammatory status through the measurements of specific biomarkers of inflammation in tracheal aspirates (in a subgroup of babies who require endotracheal intubation for mechanical ventilation when feasible);
- to assess immunogenicity through the measurement of antibodies to SP-B analogue (CHF 5736.03) and SP-C analogue (CHF 4902.03) contained in CHF 5633;
- to perform the evaluation of oxygenation status through invasive measurements [in a subgroup of babies who have an arterial (umbilical, peripheral) access, when feasible];
- to evaluate the safety profile in the two treatment groups in terms of adverse events (AEs) and adverse drug reactions (ADRs), vital signs, hematology and biochemistry values.

## 2. STUDY DESIGN

The Schedule of Assessments is presented in Appendix 1.

## 3. STUDY POPULATION

A total number of 126 (63 in each treatment group) preterm neonates with a gestational age of 24<sup>+0</sup> weeks up to 29<sup>+6</sup> weeks with RDS, will be randomized in the study. Detailed lists of inclusion and exclusion criteria are shown in Sections 4.2 and 4.3 of the CSP.

#### 4. STATISTICAL BASIS FOR SAMPLE SIZE

According to the exploratory nature of this study, no formal sample size calculation was performed. A maximum number of sixty-three randomized neonates per treatment group (126 in total) is deemed sufficient to describe the efficacy and safety of CHF5633 compared to Poractant Alfa.

Chiesi Final 1.0 CCD-5633AA1-02 18/July/2018

TP-EP.BS-WW-001-05 Effective date: 29 Jul 15

Related to: SOP-EP.BS-WW-002 

5. RANDOMIZATION

A dynamic randomization method was used to balance the treatment groups by investigational site

and gestational age group (i.e. from  $24^{+0}$  to  $26^{+6}$  weeks and from  $27^{+0}$  to  $29^{+6}$  weeks). Patients will be

centrally assigned to one of the two treatment arms on admission through an IRT system (Interactive

Response Technology, combination of voice and web response system and also referred as

IVRS/IWRS).

The IRT will allocate the patient to a certain treatment group using the Pocock and Simon

minimization algorithm (2) and assign the study medication kit number corresponding to the patients'

treatment group. IRT specification will be fully described in a specific document, created separately.

Patients will be identified by a unique number of six digits (country in first digit, investigational site

in subsequent two digits and followed by three digits with the progressive numbering of patient in

each site.

For more information refer to section 6.5 of the CSP.

6. STATISTICAL ANALYSIS CONVENTIONS

6.1 **Collected Data** 

The study schedule is enclosed as Appendix 1.

6.1.1 **Disposition data** 

The following disposition information will be recorded and listed:

Screen Date.

Enrolled Date. •

• Failed Date.

• Discontinued Date.

Reason for Failure / Early withdrawal

Completed Date.

Parental Informed Consent Date.

Chiesi Final 1.0

18/July/2018 CCD-5633AA1-02

TP-EP.BS-WW-001-05 Effective date: 29 Jul 15

#### 6.1.2 **Demographic and Background Data**

The following demographic and anthropometric information will be recorded and listed:

#### Neonate information

- Date/Time of Birth
- Gestational Age (Weeks)
- Gestational Age (Days)

GA in weeks will be derived using the following formula:

GA (weeks) + [GA(Days) / 7]

Derived value will be shown in the table. Both original and derived values will be listed.

- Sex
- Birth Weight (grams)
- Race ([blank], white, black or African American, Asian, American Indian or Alaska native, native Hawaiian or other pacific islander, other)
- Ethnicity ([blank], not Hispanic or Latino, Hispanic or Latino, not reported)
- APGAR score (Score Range: 1-10, [blank] possible)
- Any respiratory support in the delivery room? (Y/N) If yes, which method
- Chest X-Ray (CX) performed? (Y/N), performed if deemed appropriate, at screening and at Day1 24h post with
  - o Date/Time performed
  - Findings (Normal/Abnormal NCS/Abnormal CS)
  - o Specification of findings (if abnormal)
- Complications of Prematurity (NC) with
  - o Specification of complication ([Blank], Pneumothorax, Pneumopericardium, Pneumoperitoneum, Pneumomediastinum, Apnea of prematurity AOP, Necrotizing enterocolitis NEC, Patent ductus arteriosus PDA, Pneumonia, Pulmonary interstitial emphysema PIE, Pulmonary hemorrhage, Germinal matrix/Intraventricular hemorrhage (GMH/IVH,), Cerebral parenchymal hemorrhage (CPH), Neonatal jaundice, Periventricular leukomalacia (PVL,), Retinopathy of prematurity (ROP,), Bacterial sepsis and/or meningitis, Hypoglycemia, Hyperglycemia, Hypocalcemia, Hypercalcemia, Hyponatremia, Hypernatremia, Hypokalemia, Hyperkalemia)
  - o Grade of Interventricular Hemorrhage

Chiesi Final 1.0 CCD-5633AA1-02

TP-EP.BS-WW-001-05 Effective date: 29 Jul 15

Related to: SOP-EP.BS-WW-002 

18/July/2018

- Start/End Date and Time
- Ongoing (Y/N)

#### Mother information

- Mother Medical/Surgical History (only entered if clinically significant) conditions with
  - Medical Disease
  - Start/End Date
  - o Ongoing (Y/N)
- Mother Previous and Concomitant Medications with
  - Has the Subject's mother taken any Medication during the pregnancy or the delivery? (Y/N)
  - o Trade or Generic Name
  - o Start/End Date (Day, Month, Year entered separately)
  - Ongoing (Y/N)
  - o Indication
- Pregnancy History (PH).
  - Type of the delivery ([blank], spontaneous, C-section with labor, C-section without labor, emergency C-section).
  - $\circ$  Antibiotic intake during the pregnancy (Y/N).
  - Steroid intake for fetal lung maturation (Y/N) and if yes, with information how the course was ([blank], complete, incomplete).
  - Complications (verbatim, trimester ([blank], first, second, third) and treatment given or in progress(Y/N).
  - o Intrapartum complication (verbatim and treatment given (Y/N).
- Cranial Sonography (CS) with
  - Was Cranial Sonography performed? (Y/N).
  - o Date/Time of sonography (Day, Month, Year entered separately).
  - o Findings (Normal/Abnormal NCS/Abnormal CS).
  - Was Germinal Matrix Hemorrhage (GMH) / Intraventricular Hemorrhage (IVH) present? (Y/N) with district ([blank], right, left, bilateral) if answered YES.
  - o IVH Grade ([blank] or grade 1-4 possible).
  - O Was Periventricular Leukomalacia (PVL) present? (Y/N).

Chiesi Final 1.0

CCD-5633AA1-02 18/July/2018

TP-EP.BS-WW-001-05 Effective date: 29 Jul 15

Related to: SOP-EP.BS-WW-002 

Was Cerebral Parenchymal Hemorrhage present? (Y/N).

For Cranial Sonography all values measured will be listed. Screening results will be tabulated with descriptive statistics in addition.

All medical history will be coded using Version 18.0 of the Medical Dictionary for Regulatory Activities (MedDRA).

Mother previous and concomitant medication will be coded using the World Health Organization-Drug Dictionary (WHO-DD) (Version MAR2015) and will be classified by Anatomical Therapeutic Chemical (ATC) categories.

#### 6.1.3 Safety Data

## 6.1.3.1 Adverse Events and Adverse Drug Reactions

#### 6.1.3.1.1 Adverse Events

An AE is, "any untoward medical occurrence in a patient or clinical trial subject administered a medicinal (investigational or non-investigational) product and which does not necessarily have a causal relationship with this treatment." An adverse event can therefore be any unfavorable and unintended sign (including abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal (investigational or non-investigational) product, whether or not considered related to the medicinal (investigational or non-investigational) product. All AEs will be coded using the latest available version (Version 18.0) of the Medical Dictionary for Regulatory Activities (MedDRA).

A treatment-emergent adverse event (TEAE) is defined as an AE that begins or that worsens in severity during or after first intake of the study drug has been administered.

A pre-treatment AE is defined as an AE that begins before first intake of the study drug.

Any AEs with incomplete start and end dates/times will be treated as follows:

Missing onset dates (where UK and UKN indicate unknown or missing day and month respectively):

• UK-MMM-YYYY: If the month and year are different from the month and year of the first dose of study drug, assume 01-MMM-YYYY. If the month and year are the same as the first

Chiesi Final 1.0

CCD-5633AA1-02

TP-EP.BS-WW-001-05 Effective date: 29 Jul 15

Related to: SOP-EP.BS-WW-002 

dose of study drug month and year, and the end date (after any imputation) is on or after the first dose of study drug, then assume the date of the first dose of study drug. If the month and year are the same as the first dose of study drug month, and year and the end date (after any imputation) is prior to the first dose of study drug, then assume the end date for the onset date.

• DD-UK-YYYY/UK-UKN-YYYY: If the year is different from the year of first dose of study drug, assume 01-JAN-YYYY of the collected year. If the year is the same as the first dose of study drug year, and the end date (after any imputation) is on or after the first dose of study drug, then assume the date of the first dose of study drug. If the year is the same as the first dose of study drug, and the end date (after any imputation) is prior to the first dose of study drug, then assume the end date for the onset date.

Missing end dates (where UK and UKN indicate unknown or missing day and month respectively):

- UK-MMM-YYYY: Assume the last day of the month;
- DD-UKN-YYYY/UK-UKN-YYYY: Assume 31-DEC-YYYY.

Missing start/end time (where UK and UKN indicate unknown or missing day and month respectively):

- Adverse events with unknown start and/end times (but where the date is known) will be imputed with a time of 00:00 h (start) / 23:59 h (end) for the tabulations but will be shown as UK:UK in the listings (where UK = unknown). If the date is the date of treatment start will be imputed as time of start of treatment following a worst case approach.
- Adverse events with completely unknown start dates will be considered as treatmentemergent for the tabulations and will be shown as UK in the listings.

AE Duration (days) will be computed as follows:

• When both dates are completely known and AE is resolved:

Duration (days) = AE end date – AE onset date + 1

• When the AE onset date is fully known but the AE is not resolved at the end of the trial:

Duration (days) = date of completion/discontinuation – AE onset date + 1

In this case the duration will be presented as ">x days" in the listings rather than "x days"

When the AE onset date is incomplete or unknown or when the AE has resolved but with an incomplete or unknown end date, the AE duration will not be calculated, unless otherwise specified.

Chiesi Final 1.0 CCD-5633AA1-02 18/July/2018

TP-EP.BS-WW-001-05 Effective date: 29 Jul 15

Related to: SOP-EP.BS-WW-002 

AE Relative Day of Onset will be computed as follows

• Relative day of onset for pre-treatment AE:

Relative Day of Onset = AE onset date – reference date

• Relative day of onset for TEAE:

Relative Day of Onset = AE onset date - reference date + 1

where reference date is treatment date/time.

## 6.1.3.1.2 Adverse Drug Reactions

An ADR is an, "untoward and unintended response to an investigational medicinal product related to any dose administered."

For further information please refer to Section 10 of the CSP.

#### **6.1.3.1.3 Neonatal Morbidities**

The incidence of major neonatal morbidities will be monitored (for the list of neonatal morbidities and complications of prematurity see section 10.8 of the CSP). These include:

- Air leaks (pneumothorax, pneumomediastinum, pneumopericardium, pneumoperitoneum);
- anemia of prematurity;
- apnea of prematurity;
- necrotizing enterocolitis (NEC);
- patent ductus arteriosus (PDA),
- pneumonia;
- pulmonary interstitial emphysema (PIE);
- pulmonary hemorrhage;
- germinal matrix/intraventricular hemorrhage (GMH/IVH);
- cerebral parenchymal hemorrhage;
- neonatal jaundice;
- periventricular leukomalacia (PVL);
- sepsis and/or meningitis;
- Presence of the following abnormal laboratory values:

Chiesi Final 1.0

CCD-5633AA1-02 18/July/2018

TP-EP.BS-WW-001-05 Effective date: 29 Jul 15

Related to: SOP-EP.BS-WW-002 

- o hypoglycemia
- o hyperglycemia
- o hypocalcaemia
- o hypercalcemia
- o hyponatremia
- o hypernatremia
- o hypokalemia
- o hyperkalemia.

## 6.1.3.2 Clinical Laboratory Tests

The following safety laboratory parameters will be measured:

- **Biochemistry:** urea, creatinine and electrolytes (sodium, potassium, calcium, phosphorus), alanine aminotransferase (ALT), aspartate aminotransferase (AST), glucose, C-reactive protein.
- **Hematology:** full blood count (FBC).

#### 6.1.3.3 Vital Signs

The following vital signs measurements will be obtained:

- Systolic blood pressure (SBP) [mmHg];
- Diastolic blood pressure (DBP) [mmHg],
- Heart rate (bpm);
- SpO2 during administration [%].

#### 6.1.3.4 Physical Examination

Not applicable.

## 6.1.3.5 Neonatal Concomitant Medications

Any concomitant medication required for the normal care of preterm neonates will be permitted during the study. Concomitant medication will be coded using the World Health Organization-Drug

Chiesi Final 1.0

CCD-5633AA1-02

TP-EP.BS-WW-001-05 Effective date: 29 Jul 15

Related to: SOP-EP.BS-WW-002 

Dictionary (WHO-DD) (Version SEP2015) and will be classified by Anatomical Therapeutic

Chemical (ATC) categories.

6.1.3.6 Surgical/Medical Procedures

Any Surgical/ Medical Procedure required for the normal care of preterm neonates during the study

conduct will be documented with:

• Has the Subject undergone any Surgical/Medical procedures? (Y/N), if answered yes with:

o Name of the Procedure;

o Start/End Date and Time;

Adverse Event Number (assigned);

o Indication: Complication (with number and specification if other mentioned.)

and coded.

6.1.3.7 Immunogenicity Assessment

Immunogenicity assessment will be carried out in one blood sample collected prior to study treatment

administration and approximately at 5 weeks after administration (with a window from 3 to 6 weeks).

The measure of anti-SP-B and anti-SP-C antibodies will be evaluated by a titration versus a positive

control serum (GP). Further details are given in section 7.2.1 of the CSP.

6.1.4 Pharmacodynamic/Efficacy Data

6.1.4.1 Ratio of arterial oxygen saturation (SpO<sub>2</sub>/FiO<sub>2</sub>)

Ratio of arterial oxygen saturation determined by pulse oximetry and fraction of inspired oxygen

(SpO<sub>2</sub>/FiO<sub>2</sub>) will be determined in the first 7 days post-treatment (at 30 minutes, at 1, 3, 6, 12, 18, 24

hours, at Days 2, 3, 5 and 7), at Day 28±2 PNA, at discharge home and at 36 weeks PMA.

Chiesi

Final 1.0

18/July/2018

CCD-5633AA1-02

TP-EP.BS-WW-001-05 Effective date: 29 Jul 15

## 6.1.4.2 Fraction of inspired oxygen (FiO<sub>2</sub>)

FiO<sub>2</sub> will be measured in the first 7 days post treatment (at 30 minutes, at 1, 3, 6, 12, 18, 24 hours, at Days 2, 3, 5 and 7), at Day 28±2 PNA, at discharge home and at 36 weeks PMA.

#### 6.1.4.3 Arterial oxygen saturation (SpO2)

SpO<sub>2</sub> will be measured in the first 7 days post treatment (at 30 minutes, at 1, 3, 6, 12, 18, 24 hours, at Days 2, 3, 5 and 7), at Day 28±2 PNA, at discharge home and at 36 weeks PMA.

## 6.1.4.4 Respiratory Severity Score (RSS)

Respiratory Severity Score (RSS) [FiO<sub>2</sub> corrected by mean airway pressure (MAP)] will be calculated at each timepoint (i.e., at 30 minutes, at 1, 3, 6, 12, 18, 24 hours and on Day 2) as FiO<sub>2</sub> x MAP.

## 6.1.4.5 Oxygen Saturation Index (OSI)

Oxygen Saturation Index (OSI) will be calculated at each timepoint (i.e., at 30 minutes, at 1, 3, 6, 12, 18, 24 hours and on Day 2) as

FiO<sub>2</sub> x MAP x100/SpO<sub>2</sub>.

#### 6.1.4.6 Ventilator Settings

MAP (cmH<sub>2</sub>0), PIP (cmH<sub>2</sub>0) and PEEP (cmH<sub>2</sub>0) will be determined in the first 7 days post-treatment (at 30 minutes, at 1, 3, 6, 12, 18, 24 hours, at Days 2, 3, 5 and 7), at Day 28±2 PNA, at discharge home and at 36 weeks PMA.

## 6.1.4.7 Biomarkers of inflammation

CXCL8, Interleukin 1 $\beta$  (IL1 $\beta$ ), Interleukin 6 (IL6), Tumor Necrosis Factor-alpha (TNF- $\alpha$ ), myeloperoxidase (MPO) will be collected prior to study drug administration, at 24±1 hours and on day 2 (48±1 hours) in a subgroup of babies who require endotracheal intubation for mechanical ventilation, when feasible. Additionally, total proteins concentration and CXCL8/total protein, IL1 $\beta$ /total protein, IL6/total protein, TNF- $\alpha$ /total protein, MPO /total protein will also be provided.

Chiesi Final 1.0 CCD-5633AA1-02 18/July/2018

TP-EP.BS-WW-001-05 Effective date: 29 Jul 15

Related to: SOP-EP.BS-WW-002 

6.1.4.8 Mortality and BPD

Mortality

The mortality incidence at 36-week PMA and at Day 28 will be compared by treatment as for

Mortality/BPD incidence.

**RDS-Mortality** 

The RDS-associated Mortality incidence through 14 days of age will be surveyed in the

corresponding treatment group. Patients with reasons for discontinuation='RDS RELATED

DEATH" and died within 14 days of age will be considered in the counts.

Bronchopulmonary Dysplasia (BPD)

BPD is defined according to the diagnostic criteria recently proposed by the NICHD / NHLBI / ORD

Workshop [4].

The patients will be diagnosed with BPD and included in the analysis if the following applies:

Has the baby been treated with oxygen >21% for at least 28 days? ='Yes' and 'Did the patient have

a diagnosis of BPD?='Yes'.

In addition, if:

1) there is no requirement for supplemental oxygen and ventilatory support (i.e. "Is there a

requirement for supplemental oxygen?" = "No" and "Is there a requirement for ventilatory

support?"="No", BPD will classified as 'Mild'

2) if there is requirement for supplemental oxygen (i.e. 'Is there a requirement for supplemental

oxygen?" = "Yes") and oxygen value <30% then BPD will be classified as 'Moderate';

3) if there is requirement for supplemental oxygen (i.e. 'Is there a requirement for

supplemental oxygen?" = "Yes") with an oxygen value ≥30% and/or positive pressure ("Is

there a requirement for ventilatory support?"="Yes") then BPD will be classified as

'Severe'

Chiesi

Final 1.0

18/July/2018

Note: if "Is there a requirement for ventilatory support?"="Yes" but ventilatory support used is Low Flow Nasal Cannula, this shouldn't be considered as positive pressure use. Please refer to Data Review report for additional details.

## Mortality/BPD incidence

The mortality/BPD incidence at 36-week PMA will be defined as:

Incidence of neonates dead within 36-week PMA or alive at 36-week PMA with a diagnosis of BPD.

#### 6.1.4.9 Rescue medication

The percentage of patients requiring at least one rescue surfactant dose at any time during the study and within 48 hrs since last dose will be determined by treatment group. Patients with pulmonary hemorrhage during the study (displayed as adverse event with corresponding preferred term 'Pulmonary haemorrhage') will be excluded from this summary.

## 6.1.4.10 Respiratory Support and Related Duration of Ventilation (Invasive and Non-invasive)

Any respiratory Support given for the normal care of preterm neonates during the study conduct will be documented with:

- Was any respiratory support provided? (Y/N), if answered yes with:
- o Method of Ventilation (and specification if other had been mentioned);
- Start/End Date and Time.

Non-invasive ventilation will include the use of at least one of the following ventilatory supports:

- Continuous Positive Airway Pressure (CPAP)
- Bi-level Positive Airway Pressure (BiPAP)
- Nasal Intermittent Positive Pressure Ventilation (NIPPV)
- High Flow Nasal Cannula (HFNC)
- Other: Nasal Synchronized Intermittent Positive Pressure Ventilation (nSIPPV)
- Other: Nasal Synchronized Intermittent Mandatory Ventilation (nSIMV)
- Other: Nasal Intermittent Mandatory Ventilation (nIMV)
- Other: Nasal High frequency ventilation (NHFV)
- Other: Nasal Pressure Support Ventilation (NPSV)

Chiesi Final 1.0

CCD-5633AA1-02 18/July/2018

TP-EP.BS-WW-001-05 Effective date: 29 Jul 15

Related to: SOP-EP.BS-WW-002 

- Other: NIPPV-NAVAMODE
- Other: NON-INVNAVA
- Other (refer to Data Review Report for exhaustive list)

Invasive ventilation will include the use of at least one the following ventilatory support:

- High Frequency Oscillatory Ventilation (HFOV)
- HFOV/NAVAMODE
- Synchronized Intermittent Mandatory Ventilation (SIMV)
- Patient Trigger Ventilation (PTV)
- Synchronized Intermittent Positive Pressure Ventilation (SIPPV)
- Other: Intermittent Mandatory Ventilation (IMV)
- Other: A/C (assist/control)
- Other: Pressure Support Ventilation (PSV)
- Other: PPVTHRUETTUBE
- Other: SIMV/NAVA.
- Other: IMV/NAVAMODE
- Other (refer to Data Review Report for exhaustive list).

Note: Low Flow Nasal Cannula use will be summarized under "Oxygen alone".

Duration of non-invasive and invasive ventilation will be defined as total number of days when neonates received non-invasive and invasive mechanical ventilation, respectively.

Duration of ventilation (invasive and non-invasive) will be calculated as the sum of each period of received ventilation which will be calculated as ventilation end date/time minus ventilation started date/time. A review of these data will be performed during BDRM to specify whether specific adaptations of the algorithm have to be implemented.

To account for missing time in date/time when deriving duration variables, the following approaches will be used:

• Time points with unknown start and/or end times (but where the date is known) will be imputed with a time of 00:00 h or treatment administration time (1st treatment Day 1 only) for the tabulations but will be shown as NK:NK in the listings (where NK = Not Known).

Chiesi Final 1.0 CCD-5633AA1-02 18/July/2018

TP-EP.BS-WW-001-05 Effective date: 29 Jul 15

Related to: SOP-EP.BS-WW-002 

6.1.4.11 Oxygen Use and Related Duration

Any Oxygen given alone for the normal care of preterm neonates during the study conduct will be

documented with:

• Was the subject given Oxygen alone? (Y/N), if answered yes with:

Start/End Date and Time.

In addition, all the cases of "Low Flow Nasal Cannula" as reported in the ventilatory parameters

pages will be summarized under Oxygen use.

Duration of oxygen use will be calculated as sum of oxygen use/LFNC end date/time minus oxygen/

LFNC use started date/time.

To account for missing time in date/time when deriving duration variables, the following approaches

will be used:

• Time points with unknown start and/or end times (but where the date is known) will be

imputed with a time of 00:00 h or treatment administration time (1st treatment Day 1 only) for

the tabulations but will be shown as NK:NK in the listings (where NK = Not Known).

6.1.4.12 Normal breathing (i.e. at room air) patients within 24 hours

Percentage of patients with at least one reading of FiO<sub>2</sub> equal to 0.21 (i.e. at room air) within 24 hours

from first intake will be taken as estimation of normal breathing.

Additionally the median duration time to reach FiO<sub>2</sub> equal to 0.21 (normal breathing) will be

determined.

6.1.4.13 Alveolar-Arterial Gradient

The alveolar–arterial gradient (A-aO<sub>2</sub>) is used in determining the source of hypoxemia is derived on

the eCRF as difference of alveolar PO<sub>2</sub> (PaO<sub>2</sub>) and arterial PO<sub>2</sub>.

Values in the first 48 hours after the first surfactant intake (i.e., at 3, 6, 12, 18, 24 hours and on day

2) will be collected, given the challenges to placing arterial catheters in pre-term neonates.

GGD 7622 A A 1 00

Chiesi

Final 1.0

18/July/2018

6.1.4.14 Oxygenation Index

The Oxygenation Index (OI) is a calculation used in intensive care medicine to measure the fraction

of inspired oxygen (FiO<sub>2</sub>) and its usage within the body according to the following formula (lower

oxygenation index is better):

 $OI = FiO_2 * MAP / PaO_2$ .

Values in the first 48 hours after the first surfactant intake (i.e., at 3, 6, 12, 18, 24 hours and on day

2) will be collected.

**6.2 Analysis Populations** 

6.2.1 **Safety Population** 

The safety population consists of all randomized patients who took at least one dose of study

medication.

The safety population (SAF) will be used in the analysis of all safety variables.

In case of deviation between as-randomized treatment and treatment actually received, the treatment

actually received will be used in the safety analyses (i.e. an "as-treated" analysis will be performed).

6.2.2 **Intention-to-Treat Population** 

The Intention-to-Treat population (ITT) consists of all randomized patients who received at least one

dose of study medication and with at least one available evaluation of efficacy after the baseline.

The efficacy analyses will be performed based on the ITT population.

6.2.3 **Per Protocol Population** 

Considering the exploratory nature of the study, no Per Protocol (PP) analysis is planned. Hence, the need to repeat efficacy analysis on a PP population for specific efficacy parameters has been discussed

during the BDRM before database lock based on the amount and kind of major protocol violations.

Chiesi Final 1.0

18/July/2018 CCD-5633AA1-02

TP-EP.BS-WW-001-05 Effective date: 29 Jul 15

Related to: SOP-EP.BS-WW-002 

The PP Population will then consist of subjects in the ITT population with no major protocol deviations. FiO2 and SpO2/FiO2 analyses will be repeated in the PP population.

## **6.3** Statistical Analysis Methods

## 6.3.1 Listings and Descriptive Statistics

All original and derived parameters as well as population characteristics will be listed and described using summary statistics. Frequency counts (number of neonates [n] and percentages) will be made for each qualitative variable. General descriptive statistics for numeric variables will include the n (number of observed values), the mean, the standard deviation, the median, the minimum, and the maximum values. For categorical variables, the number and percent of subjects with a specific level of the variable will be presented (if not stated otherwise).

All listings will include unscheduled measurements, i.e. all measured values will be listed. Listings are to be sorted by patient number and then by visit/week/day/timepoint (where applicable).

- All listings will be presented for the randomized population. Screened neonates will be used for disposition listing.
- Randomized treatment and actual treatment will be displayed in 'Listing 16.1.7 Randomization Schedule' and misallocations, if any, will be identified with a flag (§). The actual treatment will be presented in all safety listings, while the randomized treatment will be presented in the efficacy listings.
- In case of values excluded from the analysis, specific flags will be presented.

All descriptive statistics will be presented by treatment.

## 6.3.2 Statistical Significance Level

All statistical tests will be two-sided and will be performed at the 5% level of significance, unless otherwise stated.

Chiesi Final 1.0 CCD-5633AA1-02 18/July/2018

6.3.3 Software

All statistical analyses will be performed using Statistical Analysis Software (SAS®) Version 9.2 or

later.

6.3.4 Missing Data

Generally there will be no imputation of missing data. Hence critical missing data, if any, will be

discussed during the BDRM before database lock. Decisions will be fully documented in the BDRM

Report.

6.3.5 Interim Analysis

Not applicable.

**6.3.6** Protocol Deviations

Protocol deviations detected during the study will be collected in a log file list and discussed within

(physician, Data Manager, Biostatistician, PK Scientist/Analyst and Medical Writer). The

Sponsor will evaluate the protocol deviations at the BDRM before database lock in order to estimate

their influence (major, minor) on study results and to decide whether these deviations may warrant

exclusion of a subject from the statistical analyses. Major protocol violations will be listed and

summarized by treatment.

6.3.7 Patients disposition

Reason for screening failures will be presented with a breakdown of the reasons for discontinuation.

Disposition of patients and reason for discontinuations will be presented for the randomized patients

population by treatment and overall.

Chiesi

Final 1.0

18/July/2018

6.3.8 Demographic Data

All demographic data will be presented using the ITT and safety population. Data listings and

summary tables will be provided.

6.3.9 Mother and Neonatal Concomitant Medication

Any concomitant medication given for the normal care of preterm neonates or used by the neonates'

mother during the study will be listed and displayed in a frequency table.

Tables will be presented by Anatomical Main Group (1st level of ATC), Therapeutic Subgroup (2nd

level of ATC), Chemical Subgroup (4th level of ATC) and preferred drug name, alphabetically sorted.

Code and decode will be displayed as follow:

o R, Respiratory System

o R03, Drugs for Obstructive Airway Diseases

o R03CC, Selective Beta-2-Adrenoreceptor Agonists

Salbutamol.

In the summaries, subjects experiencing more than one medication classified in the same category

(previous medications, concomitant medications) within the same anatomical main group, therapeutic

subgroups, chemical subgroup and preferred name will be counted only once.

**6.3.10** Exposure to the Investigational Medicinal Product

Drug dosing (both initial and re-dosing) information (dosing date/time, volume administered,

calculated dose administered), if available, will be presented in a listing (Appendix 16.2.5).

First and cumulative dose as well as total dose administered (mg/kg) will be summarized by

treatment. Number and percentage of neonates receiving additional study drug doses will be

summarized by treatment, overall and by number of additional doses (1 or 2).

Time since birth to first dose (h) and to each of the additional doses (h) will be summarized by

treatment.

Chiesi

Final 1.0

18/July/2018

CCD-5633AA1-02

еев зоззии о

TP-EP.BS-WW-001-05 Effective date: 29 Jul 15

6.3.11 Safety Analysis

The analysis of the safety variables will be based on the safety population.

6.3.11.1 Adverse Events

An overall summary of number and percentage of subjects with at least one treatment-emergent AEs,

SAEs, ADRs, serious ADRs and AEs leading to death will be presented by treatment. The number of

events will be also displayed.

The number and percentage of patients with at least one AE and the number of AEs will be presented

by treatment for treatment-emergent AEs, SAEs, ADRs, and AEs leading to death. The summary

results will be presented in alphabetic order for the SOC. Within each SOC, the PTs will be presented

sorted by decreasing overall frequency (not explicitly displayed).

The following listings will be produced:

• Pre-treatment AEs;

TEAEs

• ADRs;

SAEs;

TEAEs leading to death.

6.3.11.2 Clinical Safety Laboratory Tests (hematology, biochemistry)

Laboratory values (hematology, biochemistry) will be listed by neonates and study time point.

All values outside the clinical reference ranges, if available, will be flagged in the data listings. The

abnormal values will be flagged with 'L' for values below the lower limit of the clinical reference

range and 'H' for values above the upper limit of the clinical reference range and included in the

listings. Clinical significance (NCS or CS), if available, will be listed as well.

Chiesi

Final 1.0

18/July/2018

6.3.11.3 *Vital Signs* 

Vital signs data (SBP, DBP, HR, SpO<sub>2</sub> during administration) taken on Day -1 will be listed by

patient.

Descriptive statistics (n, mean, SD, median, minimum, maximum) for absolute and change from

baseline values will be presented by treatment at each time point. SpO<sub>2</sub> during administration will be

summarized as well.

Time curve of the mean change from baseline in the first week of life will be presented by treatment

group.

6.3.11.4 Immunogenicity data

The levels of antibodies in serum will be listed.

'Not reliable' immunogenicity values as defined during Blind Data Review meeting will be

flagged in the listing.

**6.3.12** Efficacy Variables

The efficacy analysis will be based on the ITT population.

The efficacy parameters will be listed by treatment and time point and will include both absolute

values and changes from baseline, where applicable.

The baseline for each of these parameters will be the last pre-dose measurement taken on Day -1

(including unscheduled measurements, if available). If no assessment exists before treatment but a

measurement is taken exactly at the same time of treatment, this will be used as baseline measurement

and mentioned for corresponding outputs. The latest won't apply to SpO2 since value collected at

time 0 is not part of efficacy assessment (See Section 9 of CSP). If measurements at date of treatment

have no time information included, it is assumed as taken before treatment time since recorded under

screening assessment.

Descriptive statistics of the absolute values and changes from baseline will also be presented.

Chiesi

Final 1.0

18/July/2018

Post-treatment unscheduled assessment won't be used in the analysis unless original assessment is not available.

#### 6.3.12.1 Statistical Analysis

#### 6.3.12.1.1 SpO<sub>2</sub>/FiO<sub>2</sub> Ratio

SpO<sub>2</sub>/FiO<sub>2</sub> will be analyzed using a linear mixed model for repeated measures (MMRM) including treatment, time point, treatment by time point interaction, investigational site and gestational age group as fixed effects and pre-dose ratio as covariate. The adjusted means in each treatment group, the adjusted mean difference between treatments and their 95% confidence intervals (CIs) at each time point and averaged over the first 24 hours will be estimated by the model. The following SAS code will be used:

```
Proc Mixed data= ... (WHERE=(time LE 24));
Class treatment time site agegrp subject;
Model var=treatment time treatment*time site agegrp baseline baseline*time / ddfm=kr;
REPEATED time / subject=subject type=UN;
Lsmeans treatment*time / PDIFF CL alpha=0.05;
Lsmeans treatment / PDIFF CL alpha=0.05; * for overall;
Estimate 'CHF5633 - Curosurf: 30 min' treatment 1 -1 treatment*time 1 0 0 0 0 0 0 -1 0 0 0 0 0 0 /CL alpha=0.05;
Estimate 'CHF5633 - Curosurf: 1 hr' treatment 1 -1 treatment*time 0 1 0 0 0 0 0 -1 0 0 0 0 0 /CL alpha=0.05;
Estimate 'CHF5633 - Curosurf: 3 hrs' treatment 1 -1 treatment*time 0 0 1 0 0 0 0 0 0 -1 0 0 0 0 /CL alpha=0.05;,
Estimate 'CHF5633 - Curosurf: 6 hrs' treatment 1 -1 treatment*time 0 0 0 1 0 0 0 0 0 0 -1 0 0 0 /CL alpha=0.05;
Estimate 'CHF5633 - Curosurf: 12 hrs' treatment 1 -1 treatment*time 0 0 0 0 1 0 0 0 0 0 0 -1 0 0 /CL alpha=0.05;
Estimate 'CHF5633 - Curosurf: 18 hrs' treatment 1 -1 treatment*time 0 0 0 0 1 0 0 0 0 0 -1 0 /CL alpha=0.05;
Estimate 'CHF5633 - Curosurf: 24 hrs' treatment 1 -1 treatment*time 0 0 0 0 0 0 1 0 0 0 0 0 -1 /CL alpha=0.05;
Estimate 'CHF5633 - Curosurf: Overall' treatment 1 -1 / CL alpha=0.05;
ods output estimates=estim lsmeans=ls means;
OUIT;
/* baseline=pre dose value, agegrp=gestational age group, time in hours */
Time profile plot of mean SpO2/FiO2 in the first 24 hours post treatment will be presented
by treatment group.
```

SpO<sub>2</sub>/FiO<sub>2</sub> will be compared between treatments at the remaining post-treatment time points (i.e., Days 2, 3, 5, 7, 28±2 PNA, at discharge home and at 36 weeks PMA) using mixed model including

Chiesi Final 1.0

CCD-5633AA1-02

TP-EP.BS-WW-001-05 Effective date: 29 Jul 15

Related to: SOP-EP.BS-WW-002 

treatment, investigational site and gestational age group as fixed effects and pre-dose ratio as covariate. These results will be displayed in a separate table.

SpO2/FiO2 summary and analyses will be repeated also in the PP population.

According to the protocol, if the discharge home coincides with 36-wks PMA assessment, data are entered once in the eCRF at 36-wks PMA. In this case, data of 36-wks PMA should be used also for discharge summary and analysis.

The following SAS code will be used:

SpO2/FiO2 will be analyzed by subgroups based on ventilator support used.

#### 6.3.12.1.2 FiO2

FiO<sub>2</sub> will be analyzed at each time point and averaged over the first 24 hours post dose using the same model used for the SpO<sub>2</sub>/FiO<sub>2</sub>. Pre-dose FiO<sub>2</sub> will be used as covariate.

Time profile plot of mean FiO<sub>2</sub> in the first 24 hours after treatment will be presented by treatment group.

FiO<sub>2</sub> will be compared between treatments at additional post-treatment time points (i.e., Days 2, 3, 5, 7, 28±2 PNA, at discharge home and at 36 weeks PMA) using linear mixed model including, treatment, investigational site and gestational age group as fixed effects and pre-dose FiO<sub>2</sub> as covariate. Same SAS code displayed in the SpO<sub>2</sub>/FiO<sub>2</sub> analysis will be used.

Chiesi Final 1.0

CCD-5633AA1-02

TP-EP.BS-WW-001-05 Effective date: 29 Jul 15

Related to: SOP-EP.BS-WW-002 

According to the protocol, if the discharge home coincides with 36-wks PMA assessment, data are

entered once in the eCRF at 36-wks PMA. In this case, data of 36-wks PMA should be used also for

discharge summary and analysis.

6.3.12.1.3 **RSS** 

RSS, calculated from ventilator settings as MAP x FiO<sub>2</sub>, will be analyzed at each time point and

averaged over the first 24 hours post study drug intake using the same model used for the SpO2/FiO2.

Time profile plot of mean RSS in the first 24 hours after treatment will be presented by treatment

group.

RSS at Day 2 will be analyzed using linear mixed model including, treatment, investigational site and

gestational age group as fixed effects.

Same SAS code displayed in the SpO<sub>2</sub>/FiO<sub>2</sub> analysis will be used.

FiO2 summary and analyses will be repeated also in the PP population.

According to the protocol, if the discharge home coincides with 36-wks PMA assessment, data are

entered once in the eCRF at 36-wks PMA. In this case, data of 36-wks PMA should be used also for

discharge summary and analysis.

6.3.12.1.4 **OSI** 

OSI, will be calculated as MAP x FiO<sub>2</sub> x 100/SpO<sub>2</sub>, will be analyzed at each time point and averaged

over the first 24 hours post study drug intake using the same model used for the SpO2/FiO2.

Same SAS code displayed in the SpO<sub>2</sub>/FiO<sub>2</sub> analysis will be used.

Time profile plot of mean OSI in the first 24 hours after treatment will be presented by treatment

group. OSI at Day 2 will be analyzed using linear mixed model including, treatment, investigational

site and gestational age group as fixed effects.

Same SAS code displayed in the SpO<sub>2</sub>/FiO<sub>2</sub> analysis will be used.

Chiesi

Final 1.0

18/July/2018

According to the protocol, if the discharge home coincides with 36-wks PMA assessment, data are entered once in the eCRF at 36-wks PMA. In this case, data of 36-wks PMA should be used also for discharge summary and analysis.

#### 6.3.12.1.5 SpO2

SpO<sub>2</sub> values as well as changes from baseline (Day -1) will be summarized by treatment group by means of descriptive statistics at each post-treatment timepoints.

According to the protocol, if the discharge home coincides with 36-wks PMA assessment, data are entered once in the eCRF at 36-wks PMA. In this case, data of 36-wks PMA should be used also for discharge summary and analysis.

#### **6.3.12.1.6** Ventilator Settings

MAP, PIP, PEEP values as well as changes from baseline (Day -1) will be summarized by treatment group by means of descriptive statistics at each post-treatment timepoints.

According to the protocol, if the discharge home coincides with 36-wks PMA assessment, data are entered once in the eCRF at 36-wks PMA. In this case, data of 36-wks PMA should be used also for discharge summary and analysis.

#### 6.3.12.1.7 BPD incidence, Mortality/BPD incidence, mortality and RDS-mortality

Mortality/BPD incidence at 36-week PMA will be compared by treatment by means of Cochran-Mantel-Haenszel (CMH), adjusting for stratification GA group. Relative risk (RR) and related 95% confidence interval will be provided using a SAS code similar to:

```
PROC FREQ DATA = ...;
WEIGHT count;
TABLE factor*treatment*response/relrisk cmh norow nocol nopercent;
RUN;
/*factor=GA group
```

Chiesi Final 1.0 CCD-5633AA1-02 18/July/2018

TP-EP.BS-WW-001-05 Effective date: 29 Jul 15

Related to: SOP-EP.BS-WW-002 

Only GA factor is included since not possible to use the combination of two factors (i.e. too few neonates by site). Please refer to DR report  $^{\star}/$ 

The incidence of BPD at 36-week PMA will be compared by treatment as for Mortality/BPD incidence. Cases not assessed at 36-week PMA visit won't be imputed. Missing cases won't be included in test statistics computation.

The mortality incidence at 36-week PMA and at Day 28 will be compared by treatment as for Mortality/BPD rate.

RDS-associated mortality incidence through 14 days of age will be compared by treatment as for Mortality/BPD rate.

#### 6.3.12.1.8 Rescue surfactant use

The percentage of patients requiring at least one rescue surfactant dose will be compared by treatment group by means of a Fisher's exact test at 5% significance interval. Odds ratio (OR) and related exact 95% CI will be also provided. Patients with pulmonary hemorrhage will be excluded from this summary.

For Fisher's exact test SAS code similar to this will be used:

```
PROC FREQ DATA = ...;
WEIGHT count;
TABLE treatment*result/measures riskdiff (CL=(WALD MN))alpha=0.05
exact fisher or / alpha=0.05;
RUN;
```

/\* option riskdiff (CL=(WALD MN)) gives the WALD CI and the CI based on inverting a score test, as suggested by Miettinen and Nurminen (1985), but can be adapted if deemed appropriate \*/

#### 6.3.12.1.9 Duration of ventilation and oxygen use

The median duration time of invasive mechanical ventilation, oxygenation and non-invasive ventilation will be compared between groups by the Mann-Whitney U-test using SAS code similar to:

Chiesi Final 1.0 CCD-5633AA1-02 18/July/2018

TP-EP.BS-WW-001-05 Effective date: 29 Jul 15

Related to: SOP-EP.BS-WW-002 

PROC NPAR1WAY DATA=... hl;

\* hl adds Hodges-Lehmann confidence interval for delta;

CLASS treatment;

VAR time;

RUN;

## 6.3.12.1.10 Normal breathing patients within 24 hours

Percentage of patients with normal breathing within 24 hours will be compared by treatment groups by means of a Fisher's exact test at 5% significance interval. Odds ratio (OR) and related exact 95% CI will be also provided.

The median duration time to reach FiO<sub>2</sub> equal to 0.21 will be compared between treatments by the Mann-Whitney U-test.

#### **6.3.12.1.11** Biomarkers of inflammation

Mean values of biomarkers of inflammation (i.e., CXCL8, IL1 $\beta$ , IL6, TNF- $\alpha$ , MPO) in the tracheal aspirates as well as change from baseline to 24 hours and on Day 2 (48 hours) will be summarized by treatment by means of descriptive statistics. Additionally, total proteins concentration and CXCL8/total protein, IL1 $\beta$ /total protein, IL6/total protein, TNF- $\alpha$ /total protein, MPO /total protein will also been included.

Biomarker values below/above the limit of quantification (BLQ/ALQ) will be imputed as follows:

- 1) BLOQ (Dil), Bad Replicate (BR) and Insufficient Volume (IV) will be considered as missing
- 2) BLOQ will be imputed by the value of low detection limit divided by 2 (Example: if the database contains a value like 0.917, 0.459 value will be imputed).
- 3) ALQ by the value of detection limit plus one unit. Since diluted values have been used the following will apply

IL6 ALQ value will be imputed with 27001 (i.e. 270\*100+1)

IL8 ALQ value will be imputed with 20201 (i.e. 202\*100+1)

MPO ALQ value will be imputed with 12400001 (i.e. 24800\*500+1)

Chiesi Final 1.0 CCD-5633AA1-02 18/July/2018

TP-EP.BS-WW-001-05 Effective date: 29 Jul 15

Related to: SOP-EP.BS-WW-002 

6.3.12.1.12 Alveolar-Arterial Gradient

The alveolar-arterial gradient (A-aO<sub>2</sub>) values as well as change from baseline in the first 48 hours

after the first surfactant intake (i.e., at 3, 6, 12, 18, 24 hours and on Day 2) will be summarized by

treatment by means of descriptive statistics.

6.3.12.1.13 Oxygenation Index

The Oxygenation Index (OI) values as well as change from baseline in the first 48 hours after the first

surfactant intake (i.e., at 3, 6, 12, 18, 24 hours and on Day 2) will be summarized by treatment by

means of descriptive statistics.

Chiesi Final 1.0 CCD-5633AA1-02 18/July/2018

TP-EP.BS-WW-001-05 Effective date: 29 Jul 15

Related to: SOP-EP.BS-WW-002 

## 7. REFERENCES

- 1. SAS® Version 9.2 of the SAS System for Personal Computers. Copyright © 2002-2003. SAS Institute Inc. SAS and all other SAS Institute Inc. product or service names are registered trademarks or trademarks of SAS Institute Inc., Cary, NC, USA.
- 2. Pocock SJ, Simon R. Sequential treatment assignment with balancing for prognostic factors in controlled clinical trials. Biometrics. 1975 Mar;31(1):103-15.
- 3. Miettinen O, Nurminen M. Comparative analysis of two rates. Statistics in Medicine 1985; 4: 213-226.
- 4. Jobe A, Bancalari E. Bronchopulmonary dysplasia. Am J Respir Crit Care Med 2001; 163:
- 5. 1723-9.

Chiesi Final 1.0 CCD-5633AA1-02 18/July/2018

TP-EP.BS-WW-001-05 Effective date: 29 Jul 15

Related to: SOP-EP.BS-WW-002 

# 8. TABLES AND LISTINGS TO BE INCLUDED IN SECTION 14 OF THE CLINICAL STUDY REPORT

All the Tables, Figures and Listings with asterisk will be included in the Key First Results package.

#### DISPOSITION AND DEMOGRAPHIC DATA

Table 14.1.1.1 Patient Disposition (All Screened)

\*Table 14.1.1.2 Patient Disposition:(All Randomized)

Table 14.1.1.5 Major Protocol Deviations (ITT population)

Table 14.1.1.6 Minor Protocol Deviations (ITT population)

\*Table 14.1.1.7 Summary of Analysis Sets (All Randomized)

\*Table 14.1.2.1 Demographic Characteristics (ITT Population)

\*Table 14.1.2.2 Demographic Characteristics (Safety Population)

Table 14.1.4.1 Chest x-Ray (Safety Population)

Table 14.1.4.2 Complications of Prematurity at Baseline (Safety Population)

Table 14.1.5.1 Mother Medical and Surgical History (Safety Population)

Table 14.1.5.2 Pregnancy History (Safety Population)

Table 14.1.6.1 Mother Previous and Concomitant Medication (Safety Population)

Table 14.1.6.2 Neonatal Concomitant Medication (Safety Population)

Table 14.1.7.1 Cranial Sonography at Screening (Safety Population)

\*Table 14.1.8.1 Treatment Exposure (Safety Population)

#### **EFFICACY DATA**

\*Table 14.2.1.1.1 Summary of Ratio of Arterial Oxygen Saturation (SpO2/FiO2) versus Time Point by Treatment (ITT Population)

Table 14.2.1.1.2 Summary of Ratio of Arterial Oxygen Saturation (SpO2/FiO2) versus Time Point by Treatment (PP Population)

Chiesi Final 1.0

CCD-5633AA1-02

TP-EP.BS-WW-001-05 Effective date: 29 Jul 15

Related to: SOP-EP.BS-WW-002 

\*Table 14.2.1.2.1 Statistical Analysis of the Arterial Oxygen Saturation (SpO2/FiO2) ratio in the First 24 hrs (ITT Population)

Table 14.2.1.2.2 Statistical Analysis of the Arterial Oxygen Saturation (SpO2/FiO2) ratio in the First 24 hrs (PP Population)

Table 14.2.1.3.1 Statistical Analysis of the Arterial Oxygen Saturation (SpO2/FiO2) Ratio – Additional Timepoints (ITT Population)

Table 14.2.1.3.2 Statistical Analysis of the Arterial Oxygen Saturation (SpO2/FiO2) Ratio – Additional Timepoints (PP Population)

\*Table 14.2.2.1.1 Summary of Fraction of inspired oxygen (FiO2, %) versus Time Point by Treatment (ITT Population)

Table 14.2.2.1.2 Summary of Fraction of inspired oxygen (FiO2, %) versus Time Point by Treatment (PP Population)

\*Table 14.2.2.2.1 Statistical Analysis of FiO2 (%) in the First 24 hrs (ITT Population)

Table 14.2.2.2.2 Statistical Analysis of FiO2 (%) in the First 24 hrs (PP Population)

Table 14.2.2.3.1 Statistical Analysis of FiO2 (%) – Additional Timepoints (ITT Population)

Table 14.2.2.3.2 Statistical Analysis of FiO2 (%) – Additional Timepoints (PP Population)

Table 14.2.2.4 Normal Breathing (i.e. at room air) Patients within 24 hours (ITT Population)

Table 14.2.3.1 Summary of Respiratory Severity Score (RSS) versus Time Point by Treatment (ITT Population)

Table 14.2.3.2 Statistical Analysis of the RSS in the First 24 hrs (ITT Population)

Table 14.2.3.3 Statistical Analysis of the RSS – Additional Timepoints (ITT Population)

Table 14.2.4.1 Summary of Oxygen Saturation Index (OSI) versus Time Point by Treatment (ITT Population)

Table 14.2.4.2 Statistical Analysis of the OSI in the First 24 hrs (ITT Population)

Table 14.2.4.3 Statistical Analysis of the OSI – Additional Timepoints (ITT Population)

Chiesi Final 1.0

CCD-5633AA1-02

TP-EP.BS-WW-001-05 Effective date: 29 Jul 15

Related to: SOP-EP.BS-WW-002 

\*Table 14.2.5 Summary of SpO2 (%) versus Time Point by Treatment (ITT Population)

Table 14.2.6 Summary of Ventilator Settings (MAP, PIP, PEEP) versus Time Point by Treatment (ITT Population)

\*Table 14.2.7 Mortality and BPD (ITT Population)

\*Table 14.2.8 Rescue Medication (ITT Population)

Table 14.2.9 Duration of Ventilation (ITT Population)

Table 14.2.10 Summary of Duration of Oxygen Use (ITT Population)

Table 14.2.11 Biomarkers (ITT Population)

Table 14.2.12 Summary of Alveolar-Arterial Gradient (A-aO2) (ITT Population)

Table 14.2.13 Summary of Oxygenation Index (OI) (ITT Population)

#### **SAFETY DATA**

*ADVERSE EVENTS* 

\*Table 14.3.1.3.1 Summary of Treatment-Emergent Adverse Events (Safety Population)

\*Table 14.3.1.3.2 Treatment-emergent Adverse Events by Treatment, System Organ Class and Preferred Term (Safety Population)

Table 14.3.1.3.3 Adverse Drug Reactions by Treatment, System Organ Class and Preferred Term (Safety Population)

\*Table 14.3.1.3.4 Serious AEs by Treatment, System Organ Class and Preferred Term (Safety Population)

Table 14.3.1.3.5 Neonatal Morbidities (Safety Population)

VITAL SIGNS

Table 14.3.4.1 Vital Signs: Actual Values and Changes from Baseline (Safety Population)

#### **FIGURES**

\*Figure 14.2.1Mean (+/-95% CI) for SpO2/FiO2 ratio by Time and Treatment

Chiesi Final 1.0 CCD-5633AA1-02 18/July/2018

CCD-5633AA1-02

TP-EP.BS-WW-001-05 Effective date: 29 Jul 15

Related to: SOP-EP.BS-WW-002 

\*Figure 14.2.2Mean (+/-95% CI) for Fraction of Inspired Oxygen by Time and Treatment

Figure 14.2.3 Mean (+/-95% CI) for Respiratory Severity Score by Time and Treatment

Figure 14.2.4 Mean (+/-95% CI) for Oxygen Saturation Index by Time and Treatment

Figure 14.2.5 Mean (+/-95% CI) for Arterial Oxygen Saturation (SpO2) by Time and Treatment

Figure 14.2.6 Mean (+/-95% CI) for MAP by Time and Treatment

Chiesi Final 1.0 CCD-5633AA1-02 18/July/2018

TP-EP.BS-WW-001-05 Effective date: 29 Jul 15

Related to: SOP-EP.BS-WW-002 

# 9. LISTINGS TO BE INCLUDED IN SECTION 16 OF THE CLINICAL STUDY REPORT

#### RANDOMIZATION SCHEDULE

Listing 16.1.7 Randomization Schedule (All Randomized)

#### SUBJECT DISPOSITION

Listing 16.2.1.1 Screening Failures (All Enrolled)

Listing 16.2.1.3. Study Discontinuation (All Randomized)

Listing 16.2.1.4 Study Visit dates (All Randomized)

Listing 16.2.1.5 Study Kits Details (All Randomized)

#### PROTOCOL DEVIATIONS

Listing 16.2.2.1: Major Protocol Deviations (All Randomized)

Listing 16.2.2.2: Minor Protocol Deviations (All Randomized)

Listing 16.2.2.3 Violation of Inclusion/Exclusion Criteria (All Randomized)

#### **ANALYSIS POPULATIONS**

Listing 16.2.3.1 Population Disposition (All Randomized)

#### **DEMOGRAPHICS AND OTHER BASELINE CHARACTERISTICS**

Listing 16.2.4.1 Demographic Characteristics (All Randomized)

Listing 16.2.4.2 Complications of Prematurity (All Randomized)

Listing 16.2.4.3 Chest X-Ray (All Randomized)

Listing 16.2.4.4 Cranial Sonography (All Randomized)

Listing 16.2.4.5.1 Mother Medical and Surgical History (All Randomized)

Listing 16.2.4.5.2 Pregnancy History (All Randomized)

Listing 16.2.4.6.1 Mother Previous and Concomitant Medication (All Randomized)

Chiesi Final 1.0

CCD-5633AA1-02

TP-EP.BS-WW-001-05 Effective date: 29 Jul 15

Related to: SOP-EP.BS-WW-002 

Listing 16.2.4.6.2 Neonatal Concomitant Medications (All Randomized)

#### COMPLIANCE AND/OR DRUG CONCENTRATION DATA

Listing 16.2.5.1 Study Medication Administration (All Randomized)

Listing 16.2.5.2 Hospital Transfer (All Randomized)

Listing 16.2.5.3 Breaking the Blind (All Randomized)

#### EFFICACY/PHARMACODYNAMIC DATA

Listing 16.2.6.1 Arterial Oxygen Saturation (SpO2), Fraction of Inspired Oxygen (FiO2), SPO2/FiO2 (All Randomized)

Listing 16.2.6.2 Ventilator Settings and Respiratory Parameters (PIP, MAP, PEEP, RSS, OSI)

Listing 16.2.6.3 A-a Oxygen Gradient and Oxygenation Index (OI)

Listing 16.2.6.4 Blood Gas Analysis (BGA) (All Randomized)

Listing 16.2.6.5 Biomarkers of Inflammation in Tracheal Aspirates (All Randomized)

Listing 16.2.6.6 Respiratory Support/Duration of Ventilation (All Randomized)

Listing 16.2.6.7 Duration of Oxygen use Alone (All Randomized)

Listing 16.2.6.8 Assessment of Mortality and BPD (All Randomized)

#### ADVERSE EVENTS

Listing 16.2.7.1 Pre Treatment Adverse Events (All Randomized)

Listing 16.2.7.2 Treatment-emergent Adverse Events (All Randomized)

Listing 16.2.7.3 Adverse Drug Reactions (All Randomized)

Listing 16.2.7.4 Serious Adverse Events (All Randomized)

Listing 16.2.7.5 Adverse Events Leading to Death (All Randomized)

Listing 16.2.7.6 Neonatal Complication of Prematurity (All Randomized)

#### LABORATORY AND OTHER SAFETY ASSESSMENTS

Chiesi Final 1.0

CCD-5633AA1-02

TP-EP.BS-WW-001-05 Effective date: 29 Jul 15

Related to: SOP-EP.BS-WW-002 

Listing 16.2.8.1 Biochemistry (All Randomized)

Listing 16.2.8.2 Hematology

Listing 16.2.8.3 Abnormal Biochemistry Values (All Randomized)

Listing 16.2.8.4 Abnormal Hematology Values

Listing 16.2.8.5 Vital Signs (All Randomized)

Listing 16.2.8.6 Immunogenicity Assessment in Serum (All Randomized)

Listing 16.2.8.7 Surgical/Medical Procedure (All Randomized)

Listing 16.2.8.8 Comments (All Randomized)

## 10. DOCUMENTATION OF STATISTICAL METHODS

Appendix 16.1.9.1: SAP and related documents

Appendix 16.1.9.2: SAS Raw output of statistical analyses

Chiesi Final 1.0 CCD-5633AA1-02 18/July/2018

TP-EP.BS-WW-001-05 Effective date: 29 Jul 15

Related to: SOP-EP.BS-WW-002 

## 11. APPENDIX

# 11.1 Study Schedule (according to protocol Amendment 1)

| | ON ADMISSION<br>PRIOR TO<br>STUDY | MINUTES/HOURS/DAYS DAYS/WEEKS | | | | | | | | | | | | | KS | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| ASSESSMENT | TREATMENT<br>WITHIN FIRST<br>24 HOURS OF<br>LIFE (Day -1) | 0 | 30'<br>(±5') | 1-h<br>(±10') | 3-h<br>(±30' | 6-h<br>(±30' | 12-h<br>(±30' | 18-h<br>(±30' | 24-h<br>(±30' | Day<br>2 | Day<br>3 | Day<br>5 | Day<br>7 | Day<br>28±2<br>PNA | Discharge<br>home | 36-<br>WEEK<br>PMA | 24-<br>month<br>clinical<br>assess. |
| Randomization/Study treatment administration | | X | | | | | | | | | | | | | | | |
| Parental Informed Consent (1) | X | | | | | | | | | | | | | | | | |
| Inclusion/Exclusion Criteria | X | | | | | | | | | | | | | | | | |
| Complications during pregnancy | X | | | | | | | | | | | | | | | | |
| Demographic data | X | | | | | | | | | | | | | | | | X |
| Apgar Score | X | | | | | | | | | | | | | | | | |
| Neonatal complications | X | | | | | | | | | | | | | | | | |
| Vital signs | X | X <sup>(+)</sup> | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Chest x-ray | X(*) | | | | | | | | X(*) | | | | | | | | |
| Cranial sonography | X(*) | | | | | | | | | | | | X<br>(**) | | (X)* | | |
| Hematology and Biochemistry | | | | | | | | | X | | | | | | | | |
| Arterial Oxygen Saturation (SpO <sub>2</sub> ) | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | |
| Ventilator settings<br>(FiO <sub>2</sub> , PIP, MAP, PEEP) (2) | X | | X | X | X | X | X | X | X | X | X | X | X | X | X | X | _ |
| A-a Oxygen gradient and OI (3) | X | | | | X | X | X | X | X | X | | | | | | | |
| Duration of oxygen alone | | | | | | | | | X | X | X | X | X | X | X | X | |
| Neonatal Concomitant Medications | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | |

Chiesi Final 1.0 CCD-5633AA1-02 18/July/2018

TP-EP.BS-WW-001-05 Effective date: 29 Jul 15

Related to: SOP-EP.BS-WW-002

| Immunogenicity assessment in serum | X | | | | | | | | | | | | | (X)*** | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Tracheal aspirates (3) | X | | | | | | | | X | X | | | | | | | |
| Assessment of BPD | | | | | | | | | | | | | | | | X | |
| Adverse Events/Adverse Drug | v | v | v | v | X | v | X | v | Х | X | X | X | v | v | v | v | |
| Reactions | Λ | Λ | Λ | Λ | Λ | Λ | Λ | Λ | Λ | Λ | Λ | Λ | Λ | Λ | Λ | Λ | |
| Bayley Scales | | | | | | | | | | | | | | | | | X |
| Health status questionnaire | | | | | | | | | | | | | | | | | X |

<sup>1.</sup> Signature of Parental Informed Consent can be obtained prior to birth or after birth;

Chiesi Final 1.0 CCD-5633AA1-02 18/July/2018

TP-EP.BS-WW-001-05 Effective date: 29 Jul 15

Related to: SOP-EP.BS-WW-002

<sup>2.</sup> PIP, MAP, PEEP to be monitored and collected until Day 7;

<sup>3.</sup> In a subgroup of babies when feasible; (X)\* Only heart rate at time 0; (X)\* When applicable, at discretion of the Investigator; (X)\*\* At least one cranial ultrasound within the first 7 days of life; (X)\*\*\* The blood sampling has to be taken with a window of 3 to 6 weeks from administration